CLINICAL TRIAL: NCT07379294
Title: Effectiveness of Using Soft Foam Dressings in Preventing Pressure Injuries During Cardiac Surger
Brief Title: Soft Foam Dressings for Pressure Injury Prevention of Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shih,Wen-Chi (Other)
Responsible Party: Sponsor-Investigator, Shih,Wen-Chi, Nurse, Fu Jen Catholic University Hospital
Organization: Fu Jen Catholic University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20250378
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Patients Undergoing Cardiac Surgery Under General Anesthesia (e.g., AVR, MVR, DVR, CABG, Type A Repair, Bentall Procedure, Heart Transplantation); Expected Surgical Duration > 4 Hours; Age ≥ 18 Years; Use of Cardiopulmonary Bypass (CPB) During Surgery; Intact Skin Preoperatively, With no Existing Pressure Injuries
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: All preventive measures will be applied after induction of anesthesia; therefore, participants will be unable to know which study group they are assigned to. In addition, the foam dressing and/or other protective measures will be removed at the end of surgery, further ensuring that participants remain unaware of their group allocation after the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): AQUACEL Foam Hydrofiber Dressing
  Interventions: Other: Intervention group
- Control Group (Other): Standard pressure injury prevention care
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — routine prevention + foam dressing applied to high-risk pressure areas (heels, sacrococcygeal area, hallux prominence
  Other Names: AQUACEL Foam Hydrofiber Dressing
  Arms: Experimental Group
Other: Control group — routine measures only (pressure-relieving pad, heel pad, towel/cotton separation, etc.)
  Other Names: Standard pressure injury prevention care
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate whether the application of soft foam dressings can reduce the occurrence of surgery-related pressure injuries among patients undergoing cardiac surgery. Specifically, this research aims to investigate differences in pressure injury outcomes before and after the intervention, and to assess the preventive effectiveness of soft foam dressings as an adjunctive skin-protection strategy.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if applying soft foam dressings (AQUACEL Foam Hydrofiber Dressing) can prevent surgery-related pressure injuries in adult patients (≥18 years) undergoing cardiac surgery under general anesthesia with cardiopulmonary bypass (CPB). The main questions it aims to answer are:

Does the use of soft foam dressings reduce the incidence of perioperative pressure injuries compared with routine skin protection measures alone? Does the intervention delay the time to pressure injury development and improve postoperative skin integrity during the first 5 postoperative days? Researchers will compare the intervention group (routine prevention + AQUACEL Foam applied to high-risk pressure areas) to the control group (routine prevention only) to see if the foam dressing intervention reduces pressure injury occurrence after cardiac surgery.

Participants will:

Be screened for eligibility and provide written informed consent Receive either routine pressure injury prevention care alone (control group) or routine care plus AQUACEL Foam dressings (intervention group) applied to pressure-prone areas (e.g., heels, sacrococcygeal region, and hallux bony prominence) Complete a demographic questionnaire (approximately 10 minutes; self-completed or assisted by the researcher)

Undergo skin assessments 6 times:

T0: during preoperative preparation T1: immediately after surgery T2-T5: once daily for 4 consecutive days after ICU transfer Have perioperative and clinical data collected from medical records (e.g., surgical duration, CPB time/temperature, laboratory values such as albumin, Hb, RBC, Hct, BUN, creatinine)

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled to undergo cardiac surgery under general anesthesia
* Use of cardiopulmonary bypass (CPB) during surgery
* Expected surgical duration greater than 4 hours
* Intact skin without pre-existing pressure injury prior to surgery

Exclusion Criteria:

* Surgical position other than supine
* Long-term bedridden status prior to hospital admission
* Altered consciousness or inability to cooperate
* History of stroke with residual limb weakness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgery-related pressure injuries | From preoperative baseline (before surgery) to postoperative day 5
  The occurrence of new pressure injuries at any anatomical site, assessed using NPIAP staging criteria. Skin assessments will be performed by trained staff at predefined perioperative time points to determine whether a pressure injury develops after surgery.

SECONDARY OUTCOMES:
Time to development of pressure injury | From end of surgery to postoperative day 5
  The time (in days) from surgery completion to the first documented occurrence of a pressure injury.
Severity stage of pressure injuries | Postoperative day 1 to postoperative day 5
  The highest NPIAP stage of any pressure injury observed during the 5 postoperative days.

OTHER OUTCOMES:
Association between intraoperative temperature maintenance and pressure injury occurrence | During surgery through postoperative day 5
  Association between intraoperative core temperature measures (e.g., lowest intraoperative temperature and/or duration of temperature below a predefined threshold) and the occurrence of new pressure injuries (NPIAP staging) during the perioperative assessment period.
Association between cardiopulmonary bypass duration and pressure injury occurrence | During surgery through postoperative day 5
  Association between cardiopulmonary bypass (CPB) time (minutes) and the occurrence of new pressure injuries (NPIAP staging) assessed from immediate postoperative period through postoperative day 5.
Association between cardiopulmonary bypass temperature and pressure injury occurrence | During surgery through postoperative day 5
  Association between CPB temperature parameters (e.g., lowest CPB temperature and temperature at CPB termination) and the occurrence of new pressure injuries (NPIAP staging) during the perioperative assessment period.